CLINICAL TRIAL: NCT05180786
Title: Error-enhanced Learning & Recovery in 2 & 3 Dimensions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, James Lanphier Patton, Co-Director, Robotics Laboratory, Arms and Hands Lab, Shirley Ryan AbilityLab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00215000
Record Dates: First submitted 2021-11-04; First posted 2022-01-06 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Cerebral Vascular Accident (CVA)/Stroke
Keywords: Upper Extremity; Rehabilitation; Arm; Robotics; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other)
  Interventions: Other: Error Fields; Other: No Error Fields
- Group 2 (Other)
  Interventions: Other: Error Fields; Other: No Error Fields

INTERVENTIONS:
Other: Error Fields — Participants will complete a reaching experiment using the robotic arm with error fields turned on.
Other: No Error Fields — Participants will complete a reaching experiment using the robotic arm with error fields turned off.

SUMMARY:
This study is being done to see how errors lead to improvement. Specifically, we are evaluating the errors stroke participants make during an upper extremity exercise program when reaching for a target using their affected arm. Once we understand the participant's reaching errors, we plan to create a customized reaching exercise according to the individual's specific error tendencies which will lead to better performance on movement ability after training.

DETAILED DESCRIPTION:
The neuroplasticity of motor re-learning is a key pathway for recovery in neurorehabilitation. One critical challenge to devising treatment plans for motor recovery is the wide variation that exists between individuals, across movement repetitions, and even within movements. Development of a learning model that looks at these factors would better relate diagnoses to treatments, providing personalization and efficiency to therapy. This proposal aims to advance rehabilitation by building a modeling framework that explores the trends and exploits a fundamental learning process - error. Our goal is to preliminarily test the direct effect of this new treatment in preparation for the randomized controlled study to come. Understanding how error leads to better performance will help us program future devices for therapy for optimal outcomes.

We are using research lab equipment at the Shirley Ryan AbilityLab (SRALab) Hospital's Robotics group. The equipment will be used to implement the reaching exercises and measure participant movement. The equipment includes:

1. Barret b.u.r.t. arm robot with Teneo forearm attachment
2. LookingGlass virtual reality display system
3. Garmin Venu Sq fitness tracking wristwatch

Study Outline:

Week 1, Visit 1: Consent, In-Person Screening, and Baseline Evaluations Participants will sign a consent form. Then, they will undergo a screening process to check if they meet all the eligibility requirements. Participants that pass the in-person screening and agree to continue with the study will complete baseline evaluations which will consistent of upper extremity outcome measures, and a preliminary reaching experiment on the b.u.r.t. robotic arm.

Weeks 2-3, Visits 2-7: Treatment Visits In the following two weeks, participants will come to the lab three times a week. They will use the robotic arm, and complete several rounds of reaching exercises while looking in the virtual reality display system. Depending on the treatment visit, participants will either take home a fitness tracker, or be asked to return it.

Week 4, Visit 8: Post-Evaluations About a week after the treatment sessions, participants will return to the lab and complete the same evaluations they completed during visit 1 to see if there is any change.

Weeks 5-8: There will be no lab visits during this time.

Week 9, Visit 9: About 5-6 weeks after the treatment visits, participants will come back for follow-up evaluations. These will be the same outcome measures completed during the baseline and post-evaluation sessions.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Chronic stroke (8+ months post stroke event) with primary motor cortex involvement
3. Hemiparesis
4. Some degree of both shoulder and elbow movement capability

Exclusion Criteria:

1. Bilateral paresis
2. Severe tactile deficits using the Two-Point Discrimination Test (participant must detect<11mm)
3. Severe proprioceptive deficits
4. Severe spasticity (Modified Ashworth >3) preventing movement
5. Aphasia, cognitive impairment, or affective dysfunction that would influence the ability to perform the experiment
6. Visual deficits, and hemispatial neglect that would prevent the subjects from seeing the targets.
7. Inability to provide an informed consent
8. severe current medical problems
9. diffuse/multiple lesion sites or multiple stroke events
10. Inability to attain and maintain testing positions
11. Botox injection to the affected upper extremity within the previous 4 months
12. Concurrent participation in upper extremity rehabilitation either as part of a research intervention protocol or a prescribed therapy
13. Participation in previous, similar robotics intervention study
14. Other neurological issues

None of the following special populations will be included in this research study:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Vulnerable Populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Perpendicular Error | 60-90 minutes

SECONDARY OUTCOMES:
Action Research Arm Test | 5-20 minutes

OTHER OUTCOMES:
Upper Extremity portion of the Fugl-Meyer | 5-20 minutes
Box and Blocks | 5-20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: James Patton, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (2):
- United States (2):
  - Shirley Ryan AbilityLab (Healthy Participants), Chicago, Illinois
  - Shirley Ryan AbilityLab, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided